CLINICAL TRIAL: NCT00748254
Title: Laser-based Photoacoustic Tomography of Human Inflammatory Arthritis
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Xueding Wang, Principal Investigator, University of Michigan
Other Study IDs: HUM00003693; R01AR060350 (NIH)
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis: Patients who have active disease affecting the joints in the hand will have Laser Based Photoacoustic Tomography (PAT), MRI, Ultrasound
  Interventions: Procedure: Laser Based Photoacoustic Tomography, MRI, Ultrasound
- Normal controls: Healthy volunteers who do not have arthritis will also have Laser Based Photoacoustic Tomography (PAT), MRI, Ultrasound on the joints of their hand
  Interventions: Procedure: laser based photoacoustic tomography, MRI, ultrasound

INTERVENTIONS:
Procedure: Laser Based Photoacoustic Tomography, MRI, Ultrasound — Healthy subjects will have scans on finger joints with any of the scanning methods described above.
  Other Names: MRI,magnetic resonance imaging; US, ultrasound; PAT, laser based photoacoustic tomography
  Groups: Rheumatoid Arthritis
Procedure: laser based photoacoustic tomography, MRI, ultrasound — Subjects with arthritis will have scans on finger joints with any of the scanning methods described above.
  Other Names: laser based photoacoustic tomography; MRI; Ultrasound
  Groups: Normal controls

SUMMARY:
The purpose of this feasibility study is to determine if a new emerging technology called photoacoustic tomography (PAT) can be adapted for use in humans for the detection of chronic rheumatoid arthritis.

DETAILED DESCRIPTION:
The objective of this proposal is to adapt photoacoustic tomography (PAT), a novel, nonionizing, noninvasive, laser-based technology, for structural and functional imaging of human peripheral joints affected by inflammatory arthritis.

Combining the advantages of both light and ultrasound scanning, PAT holds promise to present objective optical information in subsurface joint tissues with high sensitivity and high spatial resolution.

This could be of considerable help in the early detection of inflammatory joint diseases. PAT may also prove useful in further understanding the pathophysiology of these disorders and assisting with therapeutic decisions, including assessment of new pharmacological therapies.

In January 2026, the decision was made to reopen recruitment for this study to collect additional data to support future clinical trial work and funding.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older can participate in this study.
* Patients can participate in this study if they have had rheumatoid arthritis for more than 2 years and their rheumatologist has referred them to this study.
* Patients can participate as a healthy volunteer with a known history of rheumatoid arthritis.

Exclusion Criteria:

* Patients, who have electrically, magnetically or mechanically activated implants such as heart pacemaker, magnetic surgical clips, prostheses or implanted neurological stimulator.
* Pregnant patients.
* Patients who is claustrophobic.
* Patients with impaired renal function cannot participate in this study such as elevate creatinine clearance, patients on kidney dialysis etc.
* Patients with shock hypotension or unstable low blood pressure.
* Patients with Rhabdomyolysis.
* Patients who have had a contrast enhanced (with gadolinium) MRA (magnetic resonance angiography)/ or MRI within the last 3 months. (Contrast is a medication injected into a vein during a imaging examination that helps produce clearer images/pictures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are 1) people who are either healthy volunteers or have patients who have rheumatoid arthritis for more than 2 years and who have a rheumatologist who referred them to this study.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2011-12-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Photoacoustic Imaging | 10 weeks
  To determine if photoacoustic imaging (PAT) can accurately assist in the diagnosis of chronic rheumatoid arthritis, with data collected every 2 weeks for a maximum of 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Xueding Wang, Ph.D, Principal Investigator — University of Michigan
Locations (1):
- Universtity of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No